CLINICAL TRIAL: NCT02419027
Title: A Multi-center Human Study to Evaluate the Efficacy and Safety of ®GI Flora in Subjects With Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBT-GS14
Record Dates: First submitted 2015-04-13; First posted 2015-04-17 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: GI Flora
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- GI Flora (Experimental): Lactobacillus acidophilus LA1 1.312% Lactobacillus rhamnosus LR5 0.656% Lactobacillus paracasei LPC5 0.656% Bifidobacterium lactis BL3 1.312% Bifidobacterium breve BR3 1.312% Pediococcus pentosaceus SL4 1.312% Prolac-T(heat-killed L. acidophilus LA1) 24.286% Dextrose 60.000% Maltodextrin 7.154% Lemon flavor 1.000% Mg-stearate 1.000% TOTAL 100% (1.4g)%
  Interventions: Dietary Supplement: GI Flora
- placebo (Placebo Comparator): Dextrose 89.846% Maltodextrin 7.154% Lemon flavor 1.000% Mg-stearate 1.000% TOTAL 100% (1.4g)%
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: GI Flora
  Arms: GI Flora
Dietary Supplement: Placebo
  Arms: placebo

SUMMARY:
A Multi-center, Randomized, Double-blinded, Placebo-controlled Human Study to Evaluate the Efficacy and Safety of probiotic mixture(®GI Flora) in Subjects with Irritable Bowel Syndrome.

Regimen: 6 probiotics mixture >10^9/D for 8 weeks

Primary variable: visual analogue scale(VAS) assessment for abdominal pain

Secondary variable:

1. change of VAS score for abdominal pain/discomfort after 4/8-week treatment
2. daily symptom score for bloating, defecation discomfort(strain/urgency/incomplete evacuation), flatulence , feces shape, frequency of bowel movements

ELIGIBILITY:
Inclusion Criteria:

* Irritable bowel syndrome patients according to Rome III criteria
* Recurrent abdominal pain or discomfort for at least 3 days per month in the last 3 months associated with at least 2 of the following characteristics: a) improvement with defecation; b) onset associated with a change in the frequency of stool; c) onset associated with a change in form (appearance) of stool.

Exclusion Criteria:

* Intolerable or hypersensitive to GI Flora.
* Patients with active colon diverticulitis.
* History of GI surgeries except hernia repair, appendectomy, primary closure due to perforation.
* History of inflammatory bowel disease, malignancy requiring surgery or chemotherapy or radiation within 5 years.
* Patient has any condition that, in the opinion of the Investigator, would compromise the well-being of the patient or the requirements of the study.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale for abdominal pain | 8 weeks